CLINICAL TRIAL: NCT02133508
Title: Observational Trial on Long Responses in Patients With Advanced Non-Small Cell Lung Cancer Treated in Second-Line With Erlotinib
Brief Title: A Study Examining Long Response in Lung Cancer Patients Treated With Tarceva (Erlotinib)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28891
Record Dates: First submitted 2014-05-07; First posted 2014-05-08 (Estimated); Results first posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC Participants: Participants with advanced non-small cell lung cancer (NSCLC), treated in second-line with erlotinib, presenting wild-type, not tested or unknown Epidermal Growth Factor Receptor (EGFR) status, and with stable disease at the first revaluation after start of erlotinib therapy.

SUMMARY:
This multicenter, retrospective and prospective observational, cohort study will examine the effect of second-line Tarceva treatment on long response in non-small cell lung cancer (NSCLC) participants with wild type or unknown EGFR status. Participants will be observed from the start of treatment for 8 months or until death. The extension of the retrospective versus prospective observation will depend on the lag between the date of the participant enrollment and the date of beginning of erlotinib therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with stage IIIb or IV NSCLC
* Participants aged >/= 18 years
* Second-line treatment with Tarceva started before study inclusion and SD response, or CR/PR according to RECIST v1.1, lasting for at least 4 weeks

Exclusion Criteria:

* Known presence of epidermal growth factor receptor (EGFR) mutation
* Participation in a clinical trial with Tarceva during the study observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2016-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- Italy (39):
  - Policlinico Ospedaliero Ss Annunziata; U.O. Di Clinica Oncologica, Chieti, Abruzzo
  - Ospedale Civile; Divisione Di Oncologia, Pescara, Abruzzo
  - Irccs Ist. Tumori Giovanni Paolo Ii; Dipartimento Oncologia Medica, Bari, Apulia
  - Ospedale Vito Fazzi; Div. Oncoematologia, Lecce, Apulia
  - Casa Sollievo della Sofferenza - Medicina Interna, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino, Campania
  - Az. Osp. Monaldi; 1 Pneumologia Oncologica, Napoli, Campania
  - Az. Osp. Monaldi; 2 Pneumologia-Chemioterapia E Day Hospital-Pneumoncologia, Napoli, Campania
  - Azienda Ospedaliera di Rilievo Nazionale A. Cardarelli; U.O.C. di Oncologia Medica, Napoli, Campania
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale; Oncologia Medica A, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Ematologia, Modena, Emilia-Romagna
  - A.O. Universitaria Di Parma; Oncologia Medica, Parma, Emilia-Romagna
  - Ospedale Provinciale Santa Maria delle Croci, Ravenna, Emilia-Romagna
  - Arcispedale Santa Maria Nuova; Oncologia, Reggio Emilia, Emilia-Romagna
  - Policlinico Universitario Campus Biomedico; Uoc Oncologia Medica, Rome, Lazio
  - Fondazione Ptv Policlinico Tor Vergata, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini; Oncologia Medica, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini; U.O.C. Pneumologia Ad Indirizzo Oncologico 1, Rome, Lazio
  - Policlinico Umberto i di Roma; dip. Scienze Radiologiche, Oncologiche, Anatomopatologiche, Rome, Lazio
  - IFO - Istituto Regina Elena; Oncologia Medica, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - A.O. Villa Scassi; Oncologia Medica, Genoa, Liguria
  - Ospedale Valduce;U.O.S. Oncologia Ed Ematologia, Como, Lombardy
  - Az. Osp. Carlo Poma; Divisione Di Oncologia Medica, Mantova, Lombardy
  - ASST DI MONZA; Oncologia Medica, Monza, Lombardy
  - Ospedale Maggiore Della Carita; Oncologia Medica, Novara, Piedmont
  - Ospedale Oncologico A.Businco; Div. Oncologia Medica II, Cagliari, Sardinia
  - Az Ospedaliera Nuovo Garibaldi Quartiere Nesima; Oncologia Medica, Catania, Sicily
  - Casa Di Cura Di Alta Specialita La Maddalena; Dept. Oncologico Di Iii Livello, Palermo, Sicily
  - Ospedale Di Macerata; Oncologia, Macerata, The Marches
  - Ospedale Di Bolzano; Dept. Di Oncologia, Bolzano, Trentino-Alto Adige
  - Azienda Ospedaliero-Universitaria Careggi;S.C. Oncologia Medica 1, Florence, Tuscany
  - Ospedale Nuovo Della Versilia; Divisione Di Oncologia Medica, Lido di Camaiore, Tuscany
  - Ospedale Civile; Unita Operativa Di Oncologia Medica, Livorno, Tuscany
  - A.O. Universitaria Pisana-Ospedale Cisanello; Dipartimento Cardio Toracico-Pneumologia Ii, Pisa, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Seconda, Padua, Veneto
  - Ospedale Cà Foncello - Divisione di Oncologia Medica, Treviso, Veneto
  - A.O.U.I. VERONA-OSPEDALE BORGO TRENTO; ONCOLODIA MEDICA-d.O., Verona, Veneto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 172 participants were enrolled; 16 participants had protocol violations; 156 participants were eligible.
Period: Overall Study
Arm/Group | NSCLC Participants
Started | 156
Completed | 141
Not Completed | 15
Not completed — Decision of Investigator or Sponsor | 1
Not completed — Death | 12
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included eligible participants (without protocol violations).
Arm/Group | NSCLC Participants
Number analyzed (Participants) | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Stable Disease (SD) or Objective Response (Complete and Partial Response [CR + PR] According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. Objective response was defined as having a CR or PR. CR was defined as disappearance of all target and non-target lesions and no new lesions, and all pathological lymph nodes must have decreased to <10 millimeters (mm) in short axis. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. PD was defined as at least a 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and an absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: Up to 8 months
Population: All eligible participants
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Participants
Number analyzed (Participants) | 156
percentage of participants | 17.9

2. Primary Outcome: Duration of SD or Objective Response According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: The duration of SD or objective response (CR+PR) was defined as the time from first occurrence of SD or objective response to the time of PD, or death for any cause. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Objective response was defined as having a CR or PR. CR was defined as disappearance of all target and non-target lesions and no new lesions, and all pathological lymph nodes must have decreased to <10 mm in short axis. PR was defined as at least 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. PD was defined as at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and an absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: Up to 8 months
Population: All eligible participants
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Participants
Number analyzed (Participants) | 156
percentage of participants
  <2 Months | 3.8
  2-5 Months | 45.5
  5-8 Months | 28.8
  ≥8 Months | 3.8

3. Secondary Outcome: Progression-free Survival (PFS) According to RECIST v1.1
Description: PFS was defined as the time from the beginning of therapy with erlotinib to the first occurrence of disease progression, as determined by the investigator using RECIST v1.1 criteria, or death from any cause. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: Up to 8 months
Population: All eligible participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | NSCLC Participants
Number analyzed (Participants) | 156
days | 271.0 [245.0 to 304.0]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the beginning of therapy with erlotinib to death from any cause.
Time Frame: Up to 8 months
Population: All eligible participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC Participants
Number analyzed (Participants) | 156
months | NA [NA to NA] — The median value for overall survival was not estimable due to the low number of events during the observation period.

5. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is an unfavorable and unintended sign, symptom, or disease temporally associated with a clinical study, regardless of causality.
Time Frame: Up to 8 months
Population: All eligible participants
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Participants
Number analyzed (Participants) | 156
percentage of participants | 71.2

ADVERSE EVENTS:
Time Frame: Up to 8 months
Arm/Group | NSCLC Participants
Serious Adverse Events (participants affected / at risk) | 20/156
Other Adverse Events (participants affected / at risk) | 74/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC Participants (N=156)
Atrial fibrillation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Condition aggravated (General disorders) | 2
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 3
Pyrexia (General disorders) | 1
Klebsiella sepsis (Infections and infestations) | 1
Brain oedema (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Intracranial hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC Participants (N=156)
Diarrhoea (Gastrointestinal disorders) | 33
Rash (Skin and subcutaneous tissue disorders) | 62

LIMITATIONS AND CAVEATS:
Non-randomness of the recruited population; investigator-determined treatment; lack of study blinding; absence of a control group; variation in clinical settings; and evaluable sample size for assessment of the secondary objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.